CLINICAL TRIAL: NCT00936910
Title: The Use of Antifungal Lock Therapy in Intestinal Failure and Other Patients
Brief Title: Antifungal Locks to Treat Fungal-related Central Line Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bill McGhee (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Bill McGhee, Clinical Pharmacy Specialist - Transplantaton, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ambisome Locks at CHP
Record Dates: First submitted 2009-07-02; First posted 2009-07-10 (Estimated); Results first posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-09

CONDITIONS: Central Line Fungal Infections
Keywords: central line fungal infections; antifungal lock therapy; Ambisome lock therapy
MeSH Terms: interventions — Amphotericin B; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antifungal lock-treated patients (Experimental): Intestinal failure and other patients with poor IV access and central line fungal-related infections will receive intravenous systemic antifungal therapy plus the instillation of Ambisome locks into the infected catheter.
  Interventions: Drug: amphotericin B liposomal (Ambisome)

INTERVENTIONS:
Drug: amphotericin B liposomal (Ambisome) — After enrollment, antifungal therapy will be instituted consisting of both systemic and antifungal lock therapy. Systemic therapy will be amphotericin B liposomal (Ambisome) administered IV in a dose of 3-5 mg/kg/day (or other antifungal based upon standard of care) combined with antifungal lock therapy. The antifungal lock therapy consists of placing sufficient amphotericin B liposomal (Ambisome [2 mg/ml]) lock solution into the infected central venous catheter (CVC) and allowing it to dwell uninterruptedly for 8 to 12 hours per day for 10-14 days (largest CVC = 2.3 mL).
  Other Names: Ambisome

SUMMARY:
The purpose of this study is to evaluate the usefulness of antifungal lock therapy with liposomal amphotericin B (Ambisome), in combination with systemic antifungal(s), in patients with catheter-related blood stream infections with fungal organisms, whose catheter has not been removed because of the continuing critical need for central line access. The primary group of potential patients will be those with intestinal insufficiency, including post-op small bowel transplant recipients.

The recommendation of the Infectious Disease Society of America (IDSA) is to remove all catheters with fungal infections and treat systemically for 14 days after the last positive culture. However, in certain intestinal failure patients, removal of an infected line might significantly reduce or eliminate intravenous (IV) access and create a life threatening situation. Thus, the investigators' aim is to determine the usefulness of antifungal lock therapy in intestinal failure patients whose catheter has not been removed. The investigators' hope is to salvage central line catheters rather than to remove them.

DETAILED DESCRIPTION:
This is a descriptive study in intestinal failure patients with catheter-related blood stream infections (CRBSI) with fungal organisms. At present, the recommendation of the Infectious Disease Society of America (IDSA) is to remove all catheters with fungal infections and treat systemically for 14 days after the last positive culture (2). However, in intestinal failure patients who have limited IV access, removal of a line infected with Candida albicans, although recommended, might significantly reduce intravenous access and create a life threatening situation. Thus, the purpose of this study is to evaluate the use of antifungal lock therapy with liposomal amphotericin B (Ambisome) in combination with systemic antifungal therapy in patients with fungal CRBSI, whose catheter has not been removed because of the continuing critical need for central line access. The research methods are as follows:

1. Study patients will consist of in-patients hospitalized at Children's Hospital of Pittsburgh. From our intestinal failure patients followed by GI, Transplant, and Pediatric Surgical Services, we plan to enroll 25 patients. In addition, other patients with similar concerns regarding limited central venous access with catheter-related candidal bloodstream infection may also be considered for this protocol.
2. The primary group of potential patients in the study will be patients with intestinal insufficiency, including post-op small bowel recipients, whose intravenous access is limited. Thus, when a fungal CRBSI is suspected, retention of the CVC will be highly desirable. Additional subjects potentially eligible for this study would include children with cancer, those status-post bone marrow transplant, etc. who have limited central venous access and have a documented catheter-related bloodstream infection secondary to candida.
3. Once the fungal infection is established, the patient will be approached to participate in the study. The investigator(s) will fully explain the study and its benefits and risks to the patient and/or parent or guardian (if legally appointed for research) and consent and assent will be obtained.
4. Upon enrollment, antifungal therapy will be instituted consisting of both systemic and antifungal lock therapy.

   A. Ambisome at a dose of 3-5 mg/kg/day (or other appropriate antifungal based upon standard of care) will be administered intravenously B. Antifungal lock therapy with Ambisome will be administered. It consists of the placing up to 2.3 ml (based upon specific catheter types and volumes) of concentrated Ambisome into the infected CVC and allowing it to dwell uninterruptedly for 8 to 12 hours per day. The concentration of Ambisome is 2 mg/ml in sterile water (4).
5. Patients enrolled in the study will receive routine clinical care as in-patients of CHP and be monitored appropriately from an infectious disease perspective including daily blood cultures. Patients will be examined clinically for evidence of fungal-related complications (e.g., septic arthritis, endocarditis, etc.).
6. The duration of antifungal lock therapy (in addition to IV systemic antifungal therapy) will be 10-14 days.
7. After 5 days of antifungal lock therapy, the patient with a persistently positive fungal blood culture will be deemed a failure and antifungal lock therapy will be discontinued. There will be no further antifungal lock therapy permissible via this protocol and data collection for the patient will be completed as soon as possible. The primary service will be responsible for the removal of the line.
8. With successful lock therapy, additional blood cultures through the catheter will be obtained on day 5 and day 30 (or later if subject is still on systemic antifungal agents) post antifungal lock for a test of cure.

   * If a patient has a recurrence of fungal infection on culture on day 5 or day 30 post antifungal lock, pulse field gel electrophoresis will be performed on both the original and new isolate to determine if the fungal organism is the same.
   * If the organism is the same based upon electrophoretic analysis, treatment will be deemed a failure
   * If the organism is not the same, then another source for the infection will be investigated.
9. Since the standard of care would have been to remove the CVC, the primary end point of the study will be the number and percent of patients who successfully received antifungal lock therapy, i.e., those patients with at least 2 negative fungal cultures before the completion of 5 days of antifungal lock therapy and whose CVCs were not removed. Secondary endpoints will include the number of days before the cultures become negative; the development of fungal-related complications (e.g., septic arthritis, endocarditis, etc.); and the development of recurrent candidemia on day 5 and day 30 post antifungal lock therapy.
10. When medically appropriate, subjects may be discharged to complete their Ambisome® lock therapy at home. Instructions/training on how to administer lock therapy will be provided to the parents, guardian, or subject and contact with the research coordinator will be maintained while the patient is at home.
11. A patient registry will be established and offered to all subjects with central line fungal infections treated with Ambisome® locks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intestinal insufficiency and central venous access.
* Culture positive fungal-related CRBSI.
* Females of childbearing potential will be eligible for the study.
* Ambisome carries a category B Pregnancy Risk Factor. Since this is a minimal pregnancy risk category, no special precautions will be taken to determine that the patient is not pregnant.
* HIV serostatus will not be determined for the purpose of participating in this study.

Exclusion Criteria:

* Patients less than 30 days of age
* Patients greater than 21 years of age

Ages: 30 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2006-09; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill McGhee, PharmD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The entire data for all patients from the clinical trial has been published. The reference is: McGhee W, Michaels M, Martin, J, et al. Antifungal Lock Therapy with Liposomal Amphotericin B: A Prospective Trial. Journal of the Pediatric Infectious Diseases Society. 2016;5 (1): 80-4.

REFERENCES:
- [Background] Hall K, Farr B. Diagnosis and management of long-term central venous catheter infections. J Vasc Interv Radiol. 2004 Apr;15(4):327-34. doi: 10.1097/01.rvi.0000121405.46920.87. PMID 15064335
- [Background] Mermel LA, Farr BM, Sherertz RJ, Raad II, O'Grady N, Harris JS, Craven DE; Infectious Diseases Society of America; American College of Critical Care Medicine; Society for Healthcare Epidemiology of America. Guidelines for the management of intravascular catheter-related infections. Clin Infect Dis. 2001 May 1;32(9):1249-72. doi: 10.1086/320001. Epub 2001 Apr 3. No abstract available. PMID 11303260
- [Background] Raad I, Costerton W, Sabharwal U, Sacilowski M, Anaissie E, Bodey GP. Ultrastructural analysis of indwelling vascular catheters: a quantitative relationship between luminal colonization and duration of placement. J Infect Dis. 1993 Aug;168(2):400-7. doi: 10.1093/infdis/168.2.400. PMID 8335977
- [Background] Schinabeck MK, Long LA, Hossain MA, Chandra J, Mukherjee PK, Mohamed S, Ghannoum MA. Rabbit model of Candida albicans biofilm infection: liposomal amphotericin B antifungal lock therapy. Antimicrob Agents Chemother. 2004 May;48(5):1727-32. doi: 10.1128/AAC.48.5.1727-1732.2004. PMID 15105127
- [Background] Johnson DC, Johnson FL, Goldman S. Preliminary results treating persistent central venous catheter infections with the antibiotic lock technique in pediatric patients. Pediatr Infect Dis J. 1994 Oct;13(10):930-1. doi: 10.1097/00006454-199410000-00015. No abstract available. PMID 7854895
- [Background] Viale P, Petrosillo N, Signorini L, Puoti M, Carosi G. Should lock therapy always be avoided for central venous catheter-associated fungal bloodstream infections? Clin Infect Dis. 2001 Dec 1;33(11):1947-8; author reply 1949-51. doi: 10.1086/323554. No abstract available. PMID 11692310
- [Background] Kuhn DM, George T, Chandra J, Mukherjee PK, Ghannoum MA. Antifungal susceptibility of Candida biofilms: unique efficacy of amphotericin B lipid formulations and echinocandins. Antimicrob Agents Chemother. 2002 Jun;46(6):1773-80. doi: 10.1128/AAC.46.6.1773-1780.2002. PMID 12019089
- [Background] Siegman-Igra Y, Anglim AM, Shapiro DE, Adal KA, Strain BA, Farr BM. Diagnosis of vascular catheter-related bloodstream infection: a meta-analysis. J Clin Microbiol. 1997 Apr;35(4):928-36. doi: 10.1128/jcm.35.4.928-936.1997. PMID 9157155
- [Background] Blot F, Nitenberg G, Chachaty E, Raynard B, Germann N, Antoun S, Laplanche A, Brun-Buisson C, Tancrede C. Diagnosis of catheter-related bacteraemia: a prospective comparison of the time to positivity of hub-blood versus peripheral-blood cultures. Lancet. 1999 Sep 25;354(9184):1071-7. doi: 10.1016/s0140-6736(98)11134-0. PMID 10509498
- [Background] Wey SB, Mori M, Pfaller MA, Woolson RF, Wenzel RP. Hospital-acquired candidemia. The attributable mortality and excess length of stay. Arch Intern Med. 1988 Dec;148(12):2642-5. doi: 10.1001/archinte.148.12.2642. PMID 3196127
- [Background] Eppes SC, Troutman JL, Gutman LT. Outcome of treatment of candidemia in children whose central catheters were removed or retained. Pediatr Infect Dis J. 1989 Feb;8(2):99-104. PMID 2704608
- [Background] Dato VM, Dajani AS. Candidemia in children with central venous catheters: role of catheter removal and amphotericin B therapy. Pediatr Infect Dis J. 1990 May;9(5):309-14. doi: 10.1097/00006454-199005000-00002. PMID 2352815
- [Background] Nucci M, Anaissie E. Should vascular catheters be removed from all patients with candidemia? An evidence-based review. Clin Infect Dis. 2002 Mar 1;34(5):591-9. doi: 10.1086/338714. Epub 2002 Jan 24. PMID 11810600
- [Background] Castagnola E, Marazzi MG, Tacchella A, Giacchino R. Broviac catheter-related candidemia. Pediatr Infect Dis J. 2005 Aug;24(8):747. doi: 10.1097/01.inf.0000172929.23419.cb. No abstract available. PMID 16094241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were considered for enrollment if they had chronic intestinal insufficiency (including intestinal transplantation) and/or the presence of long term central venous access, and one or more positive blood cultures for yeast attributed to the central line
Groups:
- Antifungal Lock-treated Patients: This is a single arm non-randomized study consisting primarily of intestinal failure and other patients with poor IV access and central line fungal infections
  After enrollment, antifungal therapy consisted of both IV systemic and antifungal lock therapy. Systemic therapy was Ambisome (or other antifungal based upon standard of care) administered IV in a dose of 3-5 mg/kg/day combined with antifungal lock therapy. The antifungal lock therapy involved placing a catheter-specific volume (<= 2.3 ml) of concentrated Ambisome (2 mg/ml) into the infected central venous catheter (CVC) and allowing it to dwell uninterruptedly for 8 to 12 hours per day for 10-14 days.
Period: Overall Study
Arm/Group | Antifungal Lock-treated Patients
Started | 13
Completed | 10 (The primary endpt. of 2 (-) cultures within 5 d of lock therapy was met for 10 patients)
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Groups:
- Treated Patients: Patients enrolled had intestinal insufficiency (including intestinal transplantation) and/or the presence of long term central venous access, and one or more positive cultures for yeast attributed to the central line. Patients were excluded if they hypotension at the time of enrollment or need for ICU support.
Arm/Group | Treated Patients
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 7.8 [0.92 to 18.58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13
All patients with fungal catheter-related blood stream infections were potential study subjects [Number; unit: participants] | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With 2 Negative Fungal Cultures After 5 Days of Combined Systemic Antifungal and Antifungal Lock Therapy and the CVC Was Not Removed
Description: Records the number of patients with 2 negative fungal cultures after 5 days of combined systemic antifungal and antifungal lock therapy and the CVC was not removed
Time Frame: 5 days of antifungal lock treatment
Population: 13 children with long term central line venous access with positive central line fungal infections were enrolled in the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Antifungal Lock-treated Patients
Number analyzed (Participants) | 13
Participants
  number of patients with negative culture | 10
  number of patients with positive cultures | 3

2. Secondary Outcome: The Number of Days Before the Infected Central Line Culture Becomes Negative
Description: Records the mean number of days required for the cultures to become negative
Time Frame: 5 days of antifungal lock treatment
Population: All children with long term venous access with central line fungal related infections were eligible for enrollment in the trial. No one was excluded because of age, sex, or ethinicity
Measure: Mean (Full Range); unit: days
Arm/Group | Antifungal Lock-treated Patients
Number analyzed (Participants) | 13
days | 2.4 [1 to 5]

3. Secondary Outcome: The Development of Fungal-related Complications
Description: Records the number of fungal related adverse complications that occurred
Time Frame: Usually 1-28 days
Population: All children with long term central line access with fungal-related central line infections were eligible for enrollment. No one was excluded due to sex, age, race, or ethnicity
Measure: Number; unit: adverse complications
Groups:
- Antifungal Lock-treated Patients: Intestinal failure and other patients with poor IV access and central line fungal-related infections
  After enrollment, antifungal therapy will be instituted consisting of both IV systemic and antifungal lock therapy. Systemic therapy will be Ambisome administered IV in a dose of 3-5 mg/kg/day (or other antifungal based upon standard of care) combined with antifungal lock therapy. The antifungal lock therapy consists of placing up to 2.3 ml of concentrated Ambisome (2 mg/ml) into the infected central venous catheter (CVC) and allowing it to dwell uninterruptedly for 8 to 12 hours per day for 10-14 days.
Arm/Group | Antifungal Lock-treated Patients
Number analyzed (Participants) | 13
adverse complications | 0

4. Secondary Outcome: Number of Participants With Negative Cultures on Day 5 and Day 30 During the Test of Cure Period Post Antifungal Lock
Description: Records the number of participants with 2 negative cultures who completed the trial and had (-) test of cure cultures on day 5 and 30
Time Frame: 30 days
Population: All children with long term venous access with fungal related central line infections were eligible for enrollment in the trial. No one was excluded because of age, sex, race or ethnicity.
Measure: Number; unit: participants
Arm/Group | Antifungal Lock-treated Patients
Number analyzed (Participants) | 13
participants | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the course of the trial including the 30 day test of cure period. This could approach 58 days, e.g., 28 days of systemic antifungal plus 30 days until the time of the final test of cure culture
Groups:
- Antifungal Lock-treated Patients: Intestinal failure and other patients with poor IV access and central line fungal-related infections
  After enrollment, antifungal therapy will be instituted consisting of both IV systemic and antifungal lock therapy. Systemic therapy will be Ambisome administered IV in a dose of 3-5 mg/kg/day (or other antifungal based upon standard of care) combined with antifungal lock therapy. The antifungal lock therapy consists of placing up to 2.3 ml (maximum catheter size) of concentrated Ambisome (2 mg/ml) into the infected central venous catheter (CVC) and allowing it to dwell uninterruptedly for 8 to 12 hours per day for 10-14 days.
Arm/Group | Antifungal Lock-treated Patients
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No